CLINICAL TRIAL: NCT01792765
Title: Management of Ureteral Calculi Using Ultrasound Guidance: A Radiation Free Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22487 (CPHS)
Record Dates: First submitted 2013-02-11; First posted 2013-02-15 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-02

CONDITIONS: Urolithiasis
Keywords: urolithiasis; radiation free; ultrasound guidance; ureteroscopy
MeSH Terms: conditions — Urolithiasis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Arm (No Intervention): This arm will undergo ureteroscopy using conventional fluoroscopy to guide the procedure and visualize scope position, safety wire status, etc.
- Ultrasound guidance (Experimental): This arm will have intraoperative ultrasound guidance to determine safety wire position and for scope guidance.
  Interventions: Other: Ultrasound guidance

INTERVENTIONS:
Other: Ultrasound guidance — Patient will have intraoperative ultrasound .
  Other Names: Ultrasound transducer
  Arms: Ultrasound guidance

SUMMARY:
Kidney stones are very common, and can inflict a significant degree of pain and renal damage. Some stones become obstructed in the ureter, the tube that drains the kidney. In order to remove these stones, an Urologist and their team use fluoroscopic guidance to do so, this involves continuous X-ray. Flouroscopy delivers a significant dose of radiation to the patient, as well as the health care team, which has been shown to have serious health consequences. Previous studies have shown that in certain populations, like pregnant women, stones can be managed using ultrasound guidance. The investigators propose that mid and distal ureteral stones could be managed using ultrasound guidance in conjunction with conventional stone removal techniques (ureteroscopy, lithotripsy, and ureteral stent placement), in lieu of fluoroscopy, thereby minimizing radiation to healthcare staff and patients.

The investigators hypothesize that distal ureteral stones can be identified and efficiently fragmented and removed under ultrasound guidance in a safe and effective manner without the use of radiation.

DETAILED DESCRIPTION:
Patients will be enrolled and consented for this study in our Urology Clinic at Dartmouth Hitchcock Memorial Hospital and randomized prospectively to fluoroscopic versus ultrasound guided groups. A computer randomization program will be used to randomize the patient to the test or control group. Randomization will take place after they have consented to participate in the study, and the case will be booked accordingly. Consent to participate in this study will be obtained at the patient's followup appointment. At the time of the initial clinical encounter they will be provided with the consent form and information regarding the study. Once they have had the chance to look this over they will be contacted about whether they would consent to be in the study. If so, they will be randomized and the consent form signed on the morning of the procedure. Each group will consist of 25 patients. This pilot group size was determined based on feasibility of recruitment in the study period and funding availability.

All patients will receive preoperative antibiotics selected in accordance to their previous urine culture sensitivities and their respective allergies where applicable. Intraoperatively, all patients will be placed in the dorsal lithotomy position. All patients will be under general anesthesia, in both treatment arms, this is standard of care. All procedures will begin with standard cystourethroscopy, removal of the previous ureteral stent, and passage of a wire proximally into the renal pelvis. The ultrasound group will undergo intraoperative transabdominal ultrasonography by a designated ultrasonographer, and the presence of the wire, and later the ureteral stent, within the renal pelvis will be confirmed via ultrasound in all patients. The control group will undergo standard verification of wire and stent placement via fluoroscopy. Operative time as well as radiation fluoroscopy time will be recorded and compared between the two groups. At our institution, this procedure is scheduled for 140 minutes of OR time based on previous experience by our group and this individual surgeon. Stone free rate will be determined at one month post operatively with a KUB and renal ultrasound and compared between groups.

Intraoperatively, if there is concern for poor visualization, lack of progress, or technical difficulty related to the use of intraoperative ultrasound, or any other safety concerns, then this technique will be abandoned and conventional fluoroscopy will be used for this patient group. This will be apparent in the first 15 - 30 minutes of the procedure.

ELIGIBILITY:
Inclusion Criteria:

Selection criteria will include adult patients with mid and distal ureteral stones ≤8mm, and will be stented prior to presenting for their intervention. Ureteral stenting prior to ureteroscopy is the standard at Dartmouth Hitchcock Medical Center, and both the test and control group will be stented for two weeks prior to their procedure. Initial ureteral stenting will be performed using conventional fluoroscopy at the discretion of the surgeon as this may be in the acute setting and not within the scope of this trial. The mid and distal portion of the ureter refers to the segment of ureter that extends from the upper portion of the sacrum distally to the bladder.

Exclusion Criteria:

Patients will be excluded from the trial if they have had surgical resection involving the bladder or ureter, or a history of known ureteral stricture. Also, this is only for adult patients (>18yo).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-10; Primary Completion 2013-08 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Safety of ultrasound guided ureteroscopy | Day1
  We assess to see if patients had any intraoperative complications during this study, or have any post operative complications as a result of their treatment.

SECONDARY OUTCOMES:
To assess the efficacy of ultrasound guided ureteroscopy for management of distal ureteral stones. | post operatively at 4-6wks post op
  We determine if we can render patients stone free using this novel method. We also determine if this is a viable option to introduce into the OR in terms of use of operative time, which is the most expensive variable when looking at this individual urologic procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Vernon M Pais, MD, Principal Investigator — Assistant Professor at Dartmouth Hitchcock Medical Center
Locations (1):
- Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire, United States